CLINICAL TRIAL: NCT00222456
Title: Can Early Intervention Prevent Developmental Disturbances/Delays and Improve the Health of Children Born Prematurely
Brief Title: Project Early Intervention 2000
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); Norwegian Council for Mental Health (Other); Norwegian Foundation for Health and Rehabilitation (Other); The Northern Norway Health Authority (Unknown); University of Tromso (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFP 46-04; NSD-codes: MN990199; NFR-number: 132506/320; NDI 98/2638-2 TFE/- 5
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Preterm Infants; Parenting Stress
Keywords: preterm infants; early intervention; outcome; behavioral problems; parenting stress
MeSH Terms: conditions — Problem Behavior

INTERVENTIONS:
Behavioral: Sensitizing parents

SUMMARY:
The purpose of this study is to examine whether an early intervention program may improve cognitive and behavioral short and longterm outcome in preterm infants.

DETAILED DESCRIPTION:
Advances in neonatal medicine has increased the survival of infants with low birth weight. Repeatedly it has been documented an increased prevalence of psychological and medical problems in this group of children. Frequent psychological problems are intellectual disturbances, language delays, behavior problems like ADHD and learning difficulties. Usual medical problems are subnormal growth, various illnesses and neuro-developmental problems.

The high prevalence of psychological and medical risks makes this group of children target for follow-up assessments and early intervention.

The main aim of the project is to investigate whether sensitizing the parents will reduce the incidence of developmental disturbances in a group of low birth weight infants compared to a control group.

The study is carried out as a cooperation between the Departments of child- and adolescent psychiatry and pediatrics of the University Hospital in Tromsoe in Northern - Norway. 140 premature infants with birth weight less than 2000 grams are randomly distributed to an intervention and control group. In addition 70 full term infants are selected to another control.

A slightly modified version of The Vermont Intervention Program for Low Birth Weight Infants is applied to the infants in the intervention group, where the parents receive one hour of instruction from a special trained neonatal nurse one hour per day the last week before discharge (infant = 37 weeks G.A.). In addition, the parents receive four home visits during the the three first months after discharge.

Psychological and medical assessments are undertaken at ages: 36 weeks G.A., 6 months, 1, 2 3 5 years corrected for prematurity

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 2000 gram

Exclusion Criteria:

* Congenital anomalies
* Non-Norwegian speaking mother
* Triplets

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 1999-03; Study Completion 2008-09

PRIMARY OUTCOMES:
Cognitive and behavioral outcome
Parenting Stress

SECONDARY OUTCOMES:
Neurodevelopmental outcome

CONTACTS AND LOCATIONS:
Overall Officials: John Ronning, PhD, Study Chair — University of Tromsoe, Norway
Locations (1):
- Pediatric Dept. University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Landsem IP, Handegard BH, Ulvund SE, Kaaresen PI, Ronning JA. Early intervention influences positively quality of life as reported by prematurely born children at age nine and their parents; a randomized clinical trial. Health Qual Life Outcomes. 2015 Feb 22;13:25. doi: 10.1186/s12955-015-0221-9. PMID 25888838
- [Derived] Landsem IP, Handegard BH, Tunby J, Ulvund SE, Ronning JA. Early intervention program reduces stress in parents of preterms during childhood, a randomized controlled trial. Trials. 2014 Oct 4;15:387. doi: 10.1186/1745-6215-15-387. PMID 25282345
- [Derived] Hauglann L, Handegaard BH, Ulvund SE, Nordhov M, Ronning JA, Kaaresen PI. Cognitive outcome of early intervention in preterms at 7 and 9 years of age: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2015 Jan;100(1):F11-6. doi: 10.1136/archdischild-2014-306496. Epub 2014 Sep 23. PMID 25249191
- [Derived] Nordhov SM, Ronning JA, Ulvund SE, Dahl LB, Kaaresen PI. Early intervention improves behavioral outcomes for preterm infants: randomized controlled trial. Pediatrics. 2012 Jan;129(1):e9-e16. doi: 10.1542/peds.2011-0248. Epub 2011 Dec 19. PMID 22184645
- [Derived] Nordhov SM, Ronning JA, Dahl LB, Ulvund SE, Tunby J, Kaaresen PI. Early intervention improves cognitive outcomes for preterm infants: randomized controlled trial. Pediatrics. 2010 Nov;126(5):e1088-94. doi: 10.1542/peds.2010-0778. Epub 2010 Oct 11. PMID 20937650